CLINICAL TRIAL: NCT05836285
Title: The ARRC III Trial of Advanced Recovery Room Care (ARRC).
Acronym: ARRCIII
Status: Recruiting | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: Royal Adelaide Hospital (Other)
Responsible Party: Principal Investigator, Guy Ludbrook, Professor of Anaesthesia, University of Adelaide
Other Study IDs: 17557
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Post-Surgical Complication; Economic Problems
Keywords: postoperative complications; safety; health economics; quality of recovery after surgery; surgery; anaesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medium risk patients undergoing surgery: Patients undergoing surgery designated as medium risk using NSQIP risk scores
  Interventions: Other: ARRC; Other: Usual Care

INTERVENTIONS:
Other: ARRC — Eligible for ARRC and managed in ARRC unit
Other: Usual Care — Eligible for ARRC but managed elsewhere as no ARRC bed available

SUMMARY:
A postoperative high-acuity model of care (ARRC) has been shown, in a prospective cohort study of approximately 850 patients, to produce a marked improvement in patient and hospital outcomes, and hospital costs, in medium risk patients (Ludbrook G et al., JAMA Surgery 2023).

The goal of this observational study is to examine the outcomes after non-cardiac surgery of a larger group of medium risk patients receiving different forms of care -ARRC and usual ward care. The main questions it aims to answer are:

what are the outcomes for patients and hospital after the different forms of care, who receives benefit from high acuity care, what underlies the improved outcomes seen with high acuity care.

DETAILED DESCRIPTION:
Demand for essential surgery is growing, yet we face an increasingly complex casemix and budget challenges. New paradigms to deliver high value care are essential.

Advanced Recovery Room Care (ARRC) is a model of care which, at RAH, has been shown to provide substantial improvements in patient outcomes, hospital utilisation, and costs of care. Specifically, it showed when compared to usual ward care: improved Days at Home after Surgery (primary outcome), decreased in-hospital complications, and decreased mortality at 1, 3 and 12 months. This model was cost-effective compared to usual ward care: ICER of approximately -$250 per DAH

It is essential to collect high quality data on this model relevant to consumers and hospitals, in order to:

* provide a robust mechanism to ensure outcomes are maintained, and ideally improved, within our institution
* provide a mechanism to potentially allow benchmarking in the future, across institutions
* better identify which surgical subgroups receive benefit from ARRC
* provide a resource to generate and test hypotheses as to how these benefits are achieved.

To that end, the ARRC II study database is to be refined to function in essence as an ongoing registry.

This will be initially piloted at RAH, the subject of this study.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective or unplanned surgery
* Scheduled to stay in hospital at least one night after surgery
* 30-day mortality of 0.5% to 8% by the US National Safety and Quality Improvement Program risk score (NSQIP)

Exclusion Criteria:

* Undergoing cardiac surgery
* Scheduled for postoperative Intensive Care Unit management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery at Royal Adelaide Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Days at Home after surgery | 90 days after surgery
  number of days spent at usual place of residence within 90 days after surgery

SECONDARY OUTCOMES:
in-hospital complications | out to 10 days after surgery
  medical emergency response level complications
mortality | 12 months after surgery
  mortality out to 1 year after surgery
cost-effectiveness | 90 days after surgery
  cost per Day at Home improvement compared to usual care - Incremental cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ludbrook, MBBS PhD, Principal Investigator — Professor of Anaesthesia
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available to other researchers on request

REFERENCES:
- [Result] Ludbrook G, Lloyd C, Story D, Maddern G, Riedel B, Richardson I, Scott D, Louise J, Edwards S. The effect of advanced recovery room care on postoperative outcomes in moderate-risk surgical patients: a multicentre feasibility study. Anaesthesia. 2021 Apr;76(4):480-488. doi: 10.1111/anae.15260. Epub 2020 Oct 7. PMID 33027534